CLINICAL TRIAL: NCT03764579
Title: Sleep and Nutrition Intervention in Obese Children, Effects on Circadian Rhythms, Metabolic and Inflammatory Status
Brief Title: Dietary Habits and Sleep in Childhood Obesity
Acronym: INFOB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, Pilar Codoñer-Franch, Head of Pediatrics, Principal Investigator, Clinical Professor, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: University of Valencia-POG
Record Dates: First submitted 2018-11-30; First posted 2018-12-05 (Actual); Last update posted 2018-12-05 (Actual); Status verified 2018-12

CONDITIONS: Childhood Obesity; Life Style; Circadian Rhythms
MeSH Terms: conditions — Pediatric Obesity | interventions — Sleep

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sleep and diet intervention (Active Comparator)
  Interventions: Behavioral: sleep and diet intervention vs diet intervention
- diet intervention (Active Comparator)
  Interventions: Behavioral: sleep and diet intervention vs diet intervention

INTERVENTIONS:
Behavioral: sleep and diet intervention vs diet intervention — lifestyle healthy food and use Harvard plate and reduce use electronic device prior sleep.

SUMMARY:
Recruitment of obese children, classification according to sleep questionnaire and randomization in two groups to perform nutritional and sleep intervention. .

One group receives dietary intervention through recommendations. A group receives dietary and sleep intervention through recommendations. An analysis of the melatonin profile and metabolic and inflammatory status is performed by biochemistry at the beginning and end of the intervention. Determine if the intervention has improved the health of obese children.

DETAILED DESCRIPTION:
This study is carried out in children aged 7 to 14 years who are overweight or obese, in which their state and circadian rhythm variation are related by means of melatonin, biochemistry and dietary and sleep questionnaires.

An intervention is performed in which patients are classified in evening and morning. After the classification, a randomized randomization is carried out in which one group receives dietary recommendations and another group receives dietary and sleep recommendations. After 6 months of follow-up the analyzes are performed again to observe possible differences with the initial values and compare it between both groups.

ELIGIBILITY:
Inclusion Criteria:

* children between 7 and 14 years old
* overweight or obese (Body Mass Index superior to 97th percentile for age and sex).

Exclusion Criteria:

* Medicine intake,
* hyperactivity,
* infectious inflammatory processes,
* elite athletes.

Ages: 7 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes
Enrollment: 120 (Estimated)
Dates: Start 2018-11-29 (Actual); Primary Completion 2019-11-29 (Estimated); Study Completion 2020-11-29 (Estimated)

PRIMARY OUTCOMES:
Body mass index measurement, percentile for age and sex | 6 months
  comparative measurements prior after intervention

SECONDARY OUTCOMES:
melatonin concentration profile in saliva | 6 months
  comparative measurements prior after intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Pilar Codoñer Franch, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No